CLINICAL TRIAL: NCT02921984
Title: Concurrent Chemotherapy Based on Genetic Testing in Patients With High-Risk Salivary Gland Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, MD, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013HNRT01
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Salivary Gland Tumors; Head and Neck Cancer
Keywords: Salivary Gland Tumors; Head and Neck Cancer; concurrent chemotherapy; genetic testing
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Radiotherapy, Intensity-Modulated; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Docetaxel arm (Experimental): Concurrent chemotherapy with Docetaxel if genetic testing show that the patient should be sensitive to this drug.
  Interventions: Drug: Docetaxel; Radiation: Intensity-modulated radiotherapy
- Pemetrexed arm (Experimental): Concurrent chemotherapy with Pemetrexed if genetic testing show that the patient should be sensitive to this drug.
  Interventions: Radiation: Intensity-modulated radiotherapy; Drug: Pemetrexed
- Cisplatin arm (Experimental): Concurrent chemotherapy with Cisplatin if genetic testing show that the patient was nor sensitive to neither Pemetrexed nor Docetaxel
  Interventions: Radiation: Intensity-modulated radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — Docetaxel only: 80 mg/m2 on day one, every 21 days if
  Arms: Docetaxel arm
Radiation: Intensity-modulated radiotherapy — a total dose of 60-66Gy in 30-32 fractions over 6-7 weeks
Drug: Pemetrexed — Pemetrexed only: 500 mg/m2 on day one, every 21 days
  Arms: Pemetrexed arm
Drug: Cisplatin — Cisplatin only: 70 mg/m2 on day one to day three, every 21 days
  Arms: Cisplatin arm

SUMMARY:
The role of postoperative concurrent chemotherapy (CCT) has not been established for salivary gland tumors (SGTs). This prospective study was conducted to evaluate the feasibility and safety of customized CCT regimens based on the gene targets of SGTs.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of a malignant salivary gland tumor of intermediate or high-grade
2. Pathologic stage T3-4 or N1-3 or T1-2, N0 with a close (≤ 5mm) or microscopically positive surgical margin
3. Surgical resection with curative intent within 8 weeks prior to registration, with no evidence of gross tumor residual
4. No evidence of distant metastases
5. No synchronous or concurrent head and neck primary tumors
6. Karnofsky score over 60
7. Adequate organ function including the following:

   1. Absolute neutrophil count (ANC) >= 1.5 * 10^9/l
   2. Platelets count >= 100 * 10^9/l
   3. Hemoglobin >= 10 g/dl
   4. AST and ALT <= 2.5 times institutional upper limit of normal (ULN)
   5. Total bilirubin <= 1.5 times institutional ULN
   6. Creatinine clearance >= 50 ml/min
   7. Serum creatine <= 1 times ULN
8. Signed written informed consent

Exclusion Criteria:

1. Evidence of distant metastasis
2. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
3. Other previous cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
5. Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Acute toxicity profiles, graded according to the NCI CTCAE version 3.0 | up to 6 weeks

SECONDARY OUTCOMES:
Disease-free survival | 2 years
  from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Zhu, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No